CLINICAL TRIAL: NCT06190457
Title: Safety and Efficacy of Intrathecal Rituximab in 16 Children of Stage Ⅲ、ⅣNon-Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC- KY- KS-2022-141
Record Dates: First submitted 2023-06-12; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma, Non-Hodgkin; Child, Only
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: From May 2015 to December 2020, 16 children with NHL who were diagnosed in the Department of Pediatric Oncology of Sun Yat-sen Memorial Hospital of Sun Yat-sen University agreed to receive RTX intrathecal therapy and signed an informed consent form. Among them, there were 13 males and 3 females, with a male-to-female ratio of 4.33:1.00, an age of 5.1-13.1 years, and an average age of onset of 8.5 years.
  1.2 Diagnosis All children are diagnosed according to WHO lymphoma typing criteria by pathomorphological classification and immunotyping of tissue or bone marrow .
  Exclusion Criteria Patients with severe organic diseases such as heart, liver and kidney, allergic to rituximab.
  Interventions: Other: intrathecal rituximab

INTERVENTIONS:
Other: intrathecal rituximab — All children were treated with a modified NHL-BFM95 regimen for children NHL with the addition of rituximab, both intravenous and intrathecal, and rituximab intrathecal infusion is scheduled to be used simultaneously with rituximab intravenous drip. rituximab intrathecal doses are 10 mg, 15 mg, and 20 mg in increments every 3 weeks. rituximab intrathecal injection does not use methotrexate or/and cytarabine intrathecaline chemotherapy.

SUMMARY:
Objective: This study demonstrated that the efficacy and safety of intrathecal(IT) rituximab in the treatment of stage Ⅲ and Ⅳ non-Hodgkin lymphoma(NHL) in children.

Methods: We reported 16 children were histologically diagnosed as stage Ⅲ and Ⅳ NHL from September 2015 to December 2020 who received IT rituximab in Pediatric Oncology of Sun Yat-Sen Memorial Hospital were restrospectively analyzed. The clinical manifestations, central nervous system involvement,treatment plan and prognosis of patients were analyzed....

ALL patients were pathologically positive for CD20 received the modified NHL-BFM 95, while IT rituximab was arranged the day before the chemotherapy, which was simultaneously used with the intravenous infusion of rituximab. The median time of doses received by each patient was 5 times, every three weeks, with the IT dose of 10 mg,15 mg, and 20 mg in increments.

DETAILED DESCRIPTION:
Malignant lymphoma is one of the most common malignancies in children, with approximately 60 percent of cases being B-cell, non-hodgkin lymphoma (NHL) . NHL in children progresses rapidly, prone to bone marrow and central nervous system (CNS) involvement , CNS-infested NHL has a poor prognosis regardless of primary or secondary , high-intensity chemotherapy, intravenous rituximab (RTX), radiotherapy, and hematopoietic stem cell transplantation, HSCT) has limited efficacy in the treatment of these children because only a small percentage of drugs/antibodies can penetrate the blood-brain barrier . Only a limited number of intrathecal agents, primarily methotrexate, steroids, and cytarabine, have been identified that have demonstrated safety in the use of CNS-violated NHL but have not improved long-term survival in these children . Therefore, whether safe and effective intrathecal drugs can be found is the focus of the treatment and prevention of CNS-infused NHL.

Most B-cell NHL tumors express CD20 antigen in tumor tissues , RTX is a chimeric monoclonal antibody specific to B-cell CD20 antigen, and a large number of studies have confirmed that intravenous infusion of RTX has a good effect on adult and pediatric B-cell NHL . However, intravenous RTX concentrations in cerebrospinal fluid are low, ranging from 0.1 to 4.4 percent of the blood concentration, and repeated intravenous use does not increase its drug concentration in the cerebrospinal fluid . Recent small clinical studies have shown that intrathecal RTX injection is safe in adult lymphoma patients , but there are no domestic cases of intrathecal RTX use in childhood lymphoma. In this paper, 16 clinical cases of intrathecal RTX injection of stage III and IV. B-cell NHL were analyzed to explore the safety and efficacy of RTX intrathecal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of B lymphocyte NHL
2. Age≤ 18 years old
3. Normal heart and kidney function

Exclusion Criteria:

1. Heart, liver and kidney diseases
2. Allergic to rituximab

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children were diagnosed according to WHO lymphoma typing criteria by pathomorphological classification and immunophenotyping of tissues or bone marrow
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
3-year disease-free survival rate | 36 months
  DFS is the time from grouping to evidence of disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Yang Li, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
This data can be requested by sending an email to the author.